CLINICAL TRIAL: NCT06348719
Title: Medico-economic Evaluation of Robot-assisted Laparoscopy Compared With Conventional Laparoscopy in Hysterectomy for Endometrial Cancer: Multicentre Randomised Controlled Trial
Brief Title: Medico-economic Evaluation of Robot-assisted Laparoscopy Compared With Conventional Laparoscopy in Hysterectomy for Endometrial Cancer.
Acronym: ROBOT-ECO-GYN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC21_9732_ROBOT-ECO-GYN
Record Dates: First submitted 2024-03-19; First posted 2024-04-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Hysterectomies for Low- or Intermediate-risk Endometrial Carcinoma
MeSH Terms: interventions — Prospective Studies; Consent Forms; Random Allocation; Biological Products; X-Rays; Analgesics; Emergency Room Visits

STUDY DESIGN:
Intervention Model Description: As part of this project, we are proposing an original approach by combining a randomized controlled trial with a prospective observational cohort and a retrospective cohort.
  This research will therefore consist of 3 complementary studies :
  A multicenter, parallel-group, open-label, randomized controlled superiority trial (ratio 1:1) comparing two groups:
  * Group 1: laparoscopic robot-assisted hysterectomy
  * Group 2: conventional laparoscopic hysterectomy A prospective cohort based on the randomized controlled trial A retrospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Randomized study: Robot-assisted laparoscopy (Experimental): Robot-assisted laparoscopic hysterectomy
  Interventions: Procedure: Robot-assisted laparoscopy; Other: information and consent; Other: randomization; Other: Collection of socio-demographic, clinical, biological, imaging and histopathological data, treatment decision, recurrence; Other: Surgical data collection; Other: Biological data collection; Other: Collection of histological data from the surgical specimen; Other: Phone calls; Other: Pain assessment; Other: Collect of data on non-reimbursed transport; Other: Collect of everyday help; Other: Collection of the business resumption date; Other: SF36 questionnaire; Other: Questionnaire EQ5D-5L; Other: FIGO Stadium; Other: Collection of treatments (analgesics and anticoagulants up to J42, complication-related treatments, etc.); Other: Collection of adjuvant treatments; Other: Recording of any complications, emergency room visits/unscheduled consultations, additional work stoppages to the initial one
- Randomized study: conventional laparoscopy (Active Comparator): Conventional laparoscopic hysterectomy
  Interventions: Procedure: conventional laparoscopy; Other: information and consent; Other: randomization; Other: Collection of socio-demographic, clinical, biological, imaging and histopathological data, treatment decision, recurrence; Other: Surgical data collection; Other: Biological data collection; Other: Collection of histological data from the surgical specimen; Other: Phone calls; Other: Pain assessment; Other: Collect of data on non-reimbursed transport; Other: Collect of everyday help; Other: Collection of the business resumption date; Other: SF36 questionnaire; Other: Questionnaire EQ5D-5L; Other: FIGO Stadium; Other: Collection of treatments (analgesics and anticoagulants up to J42, complication-related treatments, etc.); Other: Collection of adjuvant treatments; Other: Recording of any complications, emergency room visits/unscheduled consultations, additional work stoppages to the initial one
- Prospective cohort study (Other): Prospective cohort study backed by randomized controlled trial (for patients not included in the trial due to surgeon refusal, absence of learning curve criteria for the surgeon or patient refusal, center unable to participate in the randomized study).
  Interventions: Other: Prospective cohort study; Other: information and consent; Other: Collection of socio-demographic, clinical, biological, imaging and histopathological data, treatment decision, recurrence; Other: Surgical data collection; Other: Biological data collection; Other: Collection of histological data from the surgical specimen; Other: Phone calls; Other: Pain assessment; Other: Collect of data on non-reimbursed transport; Other: Collect of everyday help; Other: Collection of the business resumption date; Other: SF36 questionnaire; Other: Questionnaire EQ5D-5L; Other: FIGO Stadium; Other: Collection of treatments (analgesics and anticoagulants up to J42, complication-related treatments, etc.); Other: Collection of adjuvant treatments; Other: Recording of any complications, emergency room visits/unscheduled consultations, additional work stoppages to the initial one
- Retrospective cohort study (Other): a retrospective cohort will be set up to provide an exhaustive overview of the approaches used for endometrial cancer, according to patient characteristics (age and BMI). It will include all patients not included in the randomized controlled trial and in the prospective cohort because the surgeon did not propose it to them, because they did not wish to be followed up for the study for 6 months, or because the surgeon considered that minimally invasive surgery was not indicated; up to a limit of 1000 inclusions.
  Interventions: Other: Retrospective cohort study; Other: information and consent; Other: Collection of data

INTERVENTIONS:
Procedure: Robot-assisted laparoscopy — The experimental procedure corresponds to robot-assisted laparoscopy.
  Arms: Randomized study: Robot-assisted laparoscopy
Procedure: conventional laparoscopy — The "control" procedure corresponds to conventional laparoscopy.
  Arms: Randomized study: conventional laparoscopy
Other: Prospective cohort study — A prospective cohort of patients will be set up to support the randomized controlled trial. Patients will be offered participation in this cohort if the center is unable to participate in the randomized trial (i.e., does not have a robot, or does not have a laparoscopic column with fluorescence), if the patient refuses randomization in the randomized controlled trial, if the surgeon refuses to randomize the patient, or if the surgeon does not meet the learning curve criteria required for robotic surgery. These patients will be followed in exactly the same way as patients included in the randomized controlled trial, once their consent has been obtained.
  Arms: Prospective cohort study
Other: Retrospective cohort study — Retrospective data collection from the medical records of all patients who underwent hysterectomy for low- or intermediate-risk endometrial cancer during the inclusion period at a participating center and who were not included in the randomized controlled trial or prospective cohort; up to a limit of 1000 inclusions. For this retrospective cohort, only data concerning initial age, BMI, histological type of cancer and surgical approach used will be collected.
  Arms: Retrospective cohort study
Other: information and consent — information and consent
Other: randomization — Randomization
  Arms: Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of socio-demographic, clinical, biological, imaging and histopathological data, treatment decision, recurrence — Collection of socio-demographic, clinical, biological, imaging and histopathological data, treatment decision, recurrence
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Surgical data collection — Surgical data collection at Day 0
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Biological data collection — Biological data collection at Day 1
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of histological data from the surgical specimen — Collection of histological data from the surgical specimen et Day 42
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Phone calls — Phone calls at Day 1, Day 3,Day 7,Day14,Day 21 , Month 3
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Pain assessment — Pain assessment at day 1 , Day 3,Day 7,Day14,Day 21 , Month 3
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collect of data on non-reimbursed transport — Collect of data on non-reimbursed transport at Day 3,Day 7,Day14,Day 21 , day 42, Month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collect of everyday help — Collect of everyday help at inclusion, Day 3,Day 7,Day14,Day 21 , day 42, Month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of the business resumption date — Collection of the business resumption date at Day 3,Day 7,Day14,Day 21 , day 42, Month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: SF36 questionnaire — SF36 questionnaire at inclusion, Day 3,Day 7,Day14,Day 21 , day 42, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Questionnaire EQ5D-5L — Questionnaire EQ5D-5L at day 1, Day 3,Day 7,Day14,Day 21 , day 42, month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: FIGO Stadium — FIGO Stadium at inclusion and Day 42
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of treatments (analgesics and anticoagulants up to J42, complication-related treatments, etc.) — Collection of treatments (analgesics and anticoagulants up to J42, complication-related treatments, etc.) at day 1, Day 3,Day 7,Day14,Day 21 , day 42, month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of adjuvant treatments — Collection of adjuvant treatments at month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Recording of any complications, emergency room visits/unscheduled consultations, additional work stoppages to the initial one — Recording of any complications, emergency room visits/unscheduled consultations, additional work stoppages to the initial one at Day 3,Day 7,Day14,Day 21 , day 42, month 3, month 6
  Arms: Prospective cohort study; Randomized study: Robot-assisted laparoscopy; Randomized study: conventional laparoscopy
Other: Collection of data — Collection of data on age, baseline, BMI, histological type of cancer and surgical approach used
  Arms: Retrospective cohort study

SUMMARY:
The standard treatment for endometrial cancer is surgery, as long as the stage of the disease and the patient's condition allow. It consists of hysterectomy (TSH) with bilateral adnexectomy. The recommended surgical approach is the minimally invasive or laparoscopic route, whose oncological safety has been demonstrated by the LAP2 study.

Since 2010 and the arrival of robotic surgery in gynaecology, the robot-assisted laparoscopic approach has gradually been used for endometrial cancer Hysterectomy.

Several studies have suggested that the cost and effectiveness of laparoscopy may vary according to the age and body mass index of the patient.

The investigators therefore hypothesise that robot-assisted laparoscopy may be more efficient than conventional laparoscopy for endometrial cancer hysterectomy in the context of an advanced learning curve in France.

The investigators therefore hypothesise that robot-assisted laparoscopy could be more efficient than conventional laparoscopy for endometrial cancer hysterectomy in the context of an advanced learning curve in France. The investigators will also test the efficiency of the surgical technique as a function of age and Body mass Index.

DETAILED DESCRIPTION:
As part of this project, the investigators are proposing an original approach by combining a randomized controlled trial with a prospective observational cohort and a retrospective cohort.

This research will therefore consist of 3 complementary studies :

A multicenter, parallel-group, open-label, randomized controlled superiority trial (ratio 1:1) comparing two groups:

* Group 1: laparoscopic robot-assisted THR
* Group 2: conventional laparoscopic STH A prospective cohort based on the randomized controlled trial A retrospective cohort Qualitative analysis of perceptions of the benefits and limitations of the surgical robot, and of the obstacles and levers to its deployment: focus groups with a sample of gynecology surgical teams from volunteer centers.

Budget impact analysis

ELIGIBILITY:
Randomized Study:

Inclusion Criteria:

* Patient with low-risk or intermediate-risk endometrial carcinoma (on pre-operative workup including histology on endometrial biopsy and pelvic and lumbo-aortic MRI) , i.e. patients with endometrioid-type endometrial adenocarcinoma cancer low-grade (grade 1 or 2) and pre-therapeutic FIGO stage I (FIGO classification 2023) on MRI.
* Indication for minimally invasive STH (laparoscopy) given by the surgeon during the pre-op consultation.
* Patient accepts the matching of pseudonymized data with the French National Health Data System (SNDS)
* Major patient.
* Patient having received information on the protocol and having signed a consent form, thus accepting randomization in the robot-assisted intervention group versus conventional laparoscopy.

Non Inclusion Criteria:

* Patient operated on by a surgeon with less than 30 cases of robotic surgery in the last year and/or with less than 50 cases of total robotic experience at the time of patient inclusion.
* Patient refuses to participate in randomized controlled trial (refuses randomization)
* The surgeon refuses the patient's participation in the randomized controlled trial (does not wish to randomize the patient).
* The center does not have a robot
* The center does not have a laparoscopic column with fluorescence
* Person under legal protection (safeguard of justice, curatorship, guardianship) or person deprived of liberty;
* Patient not affiliated to a French social security scheme
* Patient participating in another interventional trial or in Jardé off-label research that impacts study data, or in RIPH3 that impacts study data
* Pregnant or breast-feeding patient

Exclusion criteria :

* Minimally invasive procedure contraindicated by pre-operative anesthesia.
* Patient operated on by a robot other than one of the intuitive robot variants (Si, X and Xi).

Prospective cohort:

Inclusion Criteria:

* Patient with low-risk or intermediate-risk endometrial carcinoma (on pre-operative workup including histology on endometrial biopsy and pelvic and lumbo-aortic MRI) , i.e. patient with endometrioid-type endometrial adenocarcinoma cancer low-grade (grade 1 or 2) and pre-therapeutic FIGO stage I (FIGO classification 2023) on MRI .
* Indication for minimally invasive STH (laparoscopy) given by the surgeon during the pre-op consultation.
* Patient accepts the matching of pseudonymized data with the French National Health Data System (SNDS)
* Major patient.
* Patient not included in randomized controlled trial because :

  * Patient refuses to participate in randomized controlled trial (refusing randomization)
  * The surgeon refuses the patient's participation in the randomized controlled trial (does not wish to randomize the patient)
  * The center does not have a robot
  * The center does not have a laparoscopic column with fluorescence
  * The surgeon does not meet the required learning curve criteria (as a reminder: ≥ 30 cases of robotic surgery in the last year and with total robotic experience ≥ 50 procedures ) at the time of patient inclusion
* Patient has been informed about the protocol and has signed a consent form.

Non Inclusion Criteria:

* Person under legal protection (safeguard of justice, curatorship, guardianship) or person deprived of liberty;
* Patient not affiliated to a French social security scheme
* Patient participating in another interventional trial or in Jardé off-label research that impacts study data, or in RIPH3 that impacts study data
* Pregnant or breast-feeding patient

Exclusion criteria :

* Minimally invasive procedure contraindicated by pre-operative anesthesia.
* Patient operated on by a robot other than one of the intuitive robot variants (Si, X and Xi).

Retrospective cohort:

Inclusion Criteria:

* Patient with low-risk or intermediate-risk endometrial carcinoma (on pre-operative workup including histology on endometrial biopsy and pelvic and lumbo-aortic MRI) , i.e. patient with endometrioid-type endometrial adenocarcinoma cancer low-grade (grade 1 or 2) and pre-therapeutic FIGO stage I (FIGO classification 2023) on MRI).
* STH performed during the inclusion period of the randomized controlled trial and/or the prospective cohortat a participating center, regardless of the approach used, not included in the randomized controlled trial and in the prospective cohort.
* Patient not objecting to the collection and use of her data
* Patient of legal age.

Non Inclusion Criteria:

* Person under legal protection (safeguard of justice, curatorship, guardianship) or person deprived of liberty;
* Patient not affiliated to a French social security scheme

Surgeons :

Inclusion Criteria:

* Surgeon performing hysterectomy on patients included in the randomized study and/or prospective cohort
* Surgeon not objecting to the collection and use of his data

Non- inclusion Criteria:

None

First surgical assistance in the field :

Inclusion Criteria:

* First surgical assistance in the field performing hysterectomy on patients included in the randomized study and/or prospective cohort
* First surgical assistance in the field not objecting to the collection and use of his data

Non- inclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Cost-utility ratio expressed in terms of costs / QALY | 6 weeks post-operatively
  Incremental cost-utility ratio expressed in terms of costs / QALY (Quality-Adjusted Life-Year) gained with robot-assisted laparoscopy versus conventional laparoscopy in patients undergoing THR for low-risk or intermediate-risk endometrial carcinoma (i. e ; endometrioid adenocarcinoma of the endometrium grade 1 or 2 and FIGO stage 1 (FIGO 2023 classification)) in pre-therapeutic MRI) following a collective perspective at 6 weeks post-operatively.

SECONDARY OUTCOMES:
Operating time | Day 0
  Operating time
Conversion rate | month 6
  Conversion rate
Rate and nature of intraoperative complications | Day 0
  Rate and nature of intraoperative complications
Post-operative complication rate and nature at D42 (Clavien-Dindo classification) | Day 42
  Post-operative complication rate and nature at D42 (Clavien-Dindo classification)
Post-operative complication rate and nature at M6 (Clavien-Dindo classification) | Month 6
  Post-operative complication rate and nature at M6 (Clavien-Dindo classification)
Volume of intraoperative blood loss | Day 0
  Volume of intraoperative blood loss
Number of RBC, FFP, PC transfused during hospital stay | Day 3
  Number of Red Blood Cell Concentrate(s) (RBC), Fresh Frozen Plasma(s) (FFP), and Platelet Concentrate(s) (PC) transfused during hospital stay
Visual analogue scale (VAS) of pain 6h after surgery | 6 Hours after surgery
  Visual analogue evaluation (VAS) of pain 6h after surgery. Scale from 0 to 10. VAS between 1 and 3: pain of mild intensity VAS between 3 and 5: pain of moderate intensity VAS between 5 and 7: intense pain VAS greater than 7: very intense pain
Visual analogue scale (VAS) of pain 24h after surgery | 24 Hours after surgery
  Visual analogue scale (VAS) of pain 24h after surgery. Scale from 0 to 10. VAS between 1 and 3: pain of mild intensity VAS between 3 and 5: pain of moderate intensity VAS between 5 and 7: intense pain VAS greater than 7: very intense pain
Visual analogue scale (VAS) of pain D3 after surgery | Day 3
  Visual analogue scale (VAS) of pain D3 after surgery. Scale from 0 to 10. VAS between 1 and 3: pain of mild intensity VAS between 3 and 5: pain of moderate intensity VAS between 5 and 7: intense pain VAS greater than 7: very intense pain
Analgesic consumption at D1 after surgery | Day 1
  Analgesic consumption at D1 after surgery
Analgesic consumption at D3 after surgery | Day 3
  Analgesic consumption at D3 after surgery
Analgesic consumption at D7 after surgery | Day 7
  Analgesic consumption at D7 after surgery
Analgesic consumption at D14 after surgery | Day 14
  Analgesic consumption at D14 after surgery
Analgesic consumption at D21 after surgery | Day 21
  Analgesic consumption at D21 after surgery
Analgesic consumption at D42 after surgery | Day 42
  Analgesic consumption at D42 after surgery
EQ-5D-5L at inclusion after surgery | Day 0
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at inclusion after surgery. Score from 0 to 1 - 0 = deceased
  1 = in perfect health
EQ-5D-5L at D1 after surgery | Day 1
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D1 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at D3 after surgery | Day 3
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D3 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at D7 after surgery | Day 7
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D7 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at D14 after surgery | Day 14
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D14 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at D21 after surgery | Day 21
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D21 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at D42 after surgery | Day 42
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at D42 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at M3 after surgery | Month 3
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at M3 after surgery. Score from 0 to 1. 0 = deceased
  1 = in perfect health
EQ-5D-5L at M6 after surgery | Month 6
  EQ-5D-5L (Euroquol - 5 Dimensions - 5 levels) at M6 after surgery. Score from 0 to 1 0 = deceased
  1 = in perfect health
SF-36 at baseline after surgery | Day 0
  SF-36 (Short Form 36) at baseline after surgery. Score from 0 to 100. The higher the score, the better the quality of life.
SF-36 at D3 after surgery | Day 3
  SF-36 (Short Form 36) at D3 after surgery. Score from 0 to 100. The higher the score, the better the quality of life.
SF-36 at D7 after surgery | Day 7
  SF-36 (Short Form 36) at D7 after surgery. Score from 0 to 100. The higher the score, the better the quality of life.
SF-36 at D42 after surgery | Day 42
  SF-36 (Short Form 36) at D42 after surgery. Score from 0 to 100. The higher the score, the better the quality of life.
SF-36 at M6 after surgery | Month 6
  SF-36 (Short Form 36) at M6 after surgery. Score from 0 to 100. The higher the score, the better the quality of life.
Consumption of care: average length of hospital stay | Day 42
  Consumption of care between surgery and D42 and M6: average length of hospital stay in days
Consumption of care: average of number of re-hospitalizations, | Day 42
  Consumption of care between surgery and D42 and M6: average of number of re-hospitalizations
Consumption of care: average of emergency room visits | Day 42
  Consumption of care between surgery and D42 and M6: average of emergency room visits
Consumption of care: average of number of gynecologist consultations | Day 42
  Consumption of care between surgery and D42 and M6: average of number of gynecologist consultations
Consumption of care: quantity of analgesic(s) | Day 42
  Consumption of care between surgery and D42 and M6: quantity of consumption of analgesic(s) up to D42
Consumption of care: | Day 42
  Consumption of care between surgery and D42 and M6: quantity of consumption of anticoagulant(s) up to D42
Consumption of care: average of number of work stoppage(s). | Day 42
  Consumption of care between surgery and D42 and M6: average of number of work stoppage(s).
Time to initiate adjuvant treatment when indicated | Month 6
  Time to initiate adjuvant treatment when indicated (radiotherapy and/or brachytherapy and/or chemotherapy).
Vital status at 6 months | Month 6
  Patient alive or not at 6 months
Gas recovery time | Day 3
  Gas recovery time
QALYs from a collective perspective at D42 | Day 42
  Incremental cost-utility ratio expressed as costs/QALYs gained with robot-assisted laparoscopy vs. laparoscopy from a collective perspective at D42, stratified by age<or≥ at 75 and BMI<or≥ at 30 kg/m2,
QALYs from a collective perspective at M6. | Month 6
  Incremental cost-utility ratio expressed as costs/QALYs gained with robot-assisted laparoscopy versus laparoscopy from a collective perspective at M6.
Number of patients who underwent each approach | Month 36
  Number of patients who underwent each approach (laparotomy, conventional laparoscopy, robotic-assisted laparoscopy or vaginal approach) among patients operated on for low- or intermediate-risk endometrial cancer at participating centers during the inclusion period.
QALYs and average costs in relation to care consumption of patients included in the prospective cohort and in the randomized controlled trial according to the approach used and subgroups defined by age (<or> to 75 years) and BMI <or> to 30 kg/m2). | Month 36
  QALYs and average costs in relation to care consumption of patients included in the prospective cohort and in the randomized controlled trial according to the approach used and subgroups defined by age (<or≥ to 75 years) and BMI <or≥ to 30 kg/m2).
Surgical teams' perception of the benefits and limitations of robotic surgery in this indication, as well as perceived barriers and levers to the deployment of robot-assisted surgery in low- or intermediate-risk endometrial cancer. | Month 36
  Surgical teams' perception of the benefits and limitations of robotic surgery in this indication, as well as perceived barriers and levers to the deployment of robot-assisted surgery in low- or intermediate-risk endometrial cancer. Use of semi directiv interview, qualitative method
Assessment of the surgeon's physical stress during and at the end of the operation using the Borg scale | Day 0
  Assessment of the surgeon's physical stress during and at the end of the operation using the Borg scale
Assessment of the surgeon's physical stress at the end of the operation using the NASA-TLX | Day 0
  Assessment of the surgeon's physical stress at the end of the operation using the NASA-TLX
Assessment of the First surgical assistant in the operating room's physical stress at the end of the operation using the NASA-TLX | Day 0
  Assessment of the First surgical assistant in the operating room's physical stress at the end of the operation using the NASA-TLX
Assessment of the First surgical assistant in the operating room's physical stress during and at the end of the operation using the Borg-Scale | Day 0
  Assessment of the First surgical assistant in the operating room's physical stress during and at the end of the operation using the Borg-Scale.
  On a scale of 0 to 10, with 0 representing no effort and 10 representing very intense (near-maximum) effort, how would you rate your current perception of the effort required for the surgical procedure? (0: No effort; 1: Very, very easy; 2: Very easy; 3: Easy; 4: Moderate effort; 5: Average; 6: A little hard; 7: Hard; 8: Very hard; 9: Very, very hard; 10: Maximum) Legs; Back; Neck; Left shoulder; Right shoulder; Left forearm; Right forearm; Left wrist; Right wrist; Left hand; Right hand; Left fingers; Right fingers
Total annual costs of the foreseeable spread of robot-assisted surgery | Month 36
  Total annual costs of the foreseeable spread of robot-assisted surgery for low-risk or intermediate-risk endometrial cancer and of alternative management, with gradual generalization over a 5-year period, based on the outlook for the French healthcare system.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU de Lille, Hôpital Jeanne de Flandre, Lille
  - CHU LIMOGES, Hôpital Mère-Enfant, Limoges
  - Hôpital Lariboisière/Hôpital Saint Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat, Paris
  - Hôpital Tenon AP-HP, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Lyon Sud - Hospices Civils de Lyon, Pierre-Bénite
  - Hôpital privé des côtes d'Armor, Plérin
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHU de Tours - Hôpital Bretonneau, Tours